CLINICAL TRIAL: NCT00713713
Title: Hemodynamic Impact of Low and High Tidal Volume Mechanical Ventilation in Acute Lung Injury (ALI)/Acute Respiratory Distress Syndrome (ARDS) Patients
Brief Title: Effect of Different Ventilatory Strategies on Cardiac Function in Patients With Acute Respiratory Failure
Acronym: VITALI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Natalini Giuseppe, FPoliambulanza
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: FP-TIP-02
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Respiratory Distress Syndrome
Keywords: Respiratory Distress Syndrome, Adult; Tidal volume; cardiac output; Respiration, Artificial; Protective ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration | interventions — Respiration, Artificial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Two different tidal volumes (6 and 12 ml.kg-1 of ideal weight) are alternatively delivered to patients 30 minutes each one. The order of the two tidal volumes is randomized. Between the two study tidal volumes, patient returns for 30 minutes to the tidal volume used before the study recruitment.
  Interventions: Procedure: Mechanical ventilation with low and high tidal volume

INTERVENTIONS:
Procedure: Mechanical ventilation with low and high tidal volume — Tidal volume of 6 or 12 ml.kg-1, calculated on ideal body weight

SUMMARY:
Mechanical ventilation with low tidal volume (about 6 ml.kg-1) reduces mortality in ALI/ARDS patients respect to high tidal volume ventilation (about 12 ml.kg-1).

This finding is usually explained by alveolar tidal overdistension associated to high tidal volume. Stretch-induced lung injury may trigger a cytokine-mediated inflammatory response. This may contribute to the development of systemic inflammatory response and multiple system organ failure and death.

High tidal volume strategies might affect organ function by pathways not mediated by inflammatory response.

It is well recognized the inverse relationship between tidal volume and cardiac output during mechanical ventilation. Nevertheless there are no clinical studies about cardiac output changes induced by low (6 ml.kg-1) and high tidal volume (12 ml.kg-1) in ALI/ARDS patients.

The study hypothesis is that high tidal volume ventilation reduces cardiac output in ALI/ARDS patients respect to low tidal volume strategy. Thereafter reduced hemodynamic impact could explain beneficial effect of low respect to high tidal volume ventilation.

If study hypothesis is confirmed, other studies should define the main cause of mortality reduction related to low tidal volume strategies and if appropriate hemodynamic monitoring and support should be required when low tidal volume strategies are harmful (i.e. traumatic brain injury).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ARDS/ALI

Exclusion Criteria:

* mean arterial pressure lower than 65 mmHg
* beginning or change of vasoactive agents infusion rate in the last 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
cardiac index | after 30 minutes of mechanical ventilation with tidal volume of 6 or 12 ml.kg-1

SECONDARY OUTCOMES:
oxygen delivery | after 30 minutes of mechanical ventilation with tidal volume of 6 or 12 ml.kg-1
oxygen consumption | after 30 minutes of mechanical ventilation with tidal volume of 6 or 12 ml.kg-1
mixed venous saturation | after 30 minutes of mechanical ventilation with tidal volume of 6 or 12 ml.kg-1
relationship between partitioned elastance (lung and chest wall) and cardiac index difference between ventilation with tidal volume 6 and 12 ml.kg-1 | after 30 minutes of mechanical ventilation with tidal volume of 6 or 12 ml.kg-1
abdominal perfusion pressure (mean arterial pressure minus abdominal pressure) | after 30 minutes of mechanical ventilation with tidal volume of 6 or 12 ml.kg-1

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Natalini, MD, Principal Investigator — Fondazione Poliambulanza Istituto Ospedaliero
Locations (1):
- Intensive Care Unit, Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Italy

REFERENCES:
- [Derived] Natalini G, Minelli C, Rosano A, Ferretti P, Militano CR, De Feo C, Bernardini A. Cardiac index and oxygen delivery during low and high tidal volume ventilation strategies in patients with acute respiratory distress syndrome: a crossover randomized clinical trial. Crit Care. 2013 Jul 23;17(4):R146. doi: 10.1186/cc12825. PMID 23880084